CLINICAL TRIAL: NCT03713268
Title: Intraoperative OCT Guidance of Intraocular Surger
Brief Title: Intraoperative OCT Guidance of Intraocular Surgery II
Acronym: MIOCT
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00100437; U01EY028079 (NIH)
Record Dates: First submitted 2018-10-15; First posted 2018-10-19 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Macular Holes; Epiretinal Membrane; Diabetic Retinopathy; Retinal Detachment; Retinal Disease; Preretinal Fibrosis; Cataract; Ocular Tumor; Strabismus; Healthy
Keywords: Microscope Integrated optical coherence tomography; MIOCT; OCT Angiography; OCTA
MeSH Terms: conditions — Retinal Perforations; Epiretinal Membrane; Diabetic Retinopathy; Retinal Detachment; Retinal Diseases; Cataract; Eye Neoplasms; Strabismus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Healthy (ocular health) participants: Adult subjects with normal, ocular health will be enrolled to evaluate and obtain multiple images from the microscope integrated optical coherence tomography system for reproducibility testing in humans, provide feedback to engineers, and verify that the system functions to produce high quality images of the desired areas of the eye after ex vivo development before surgical use.
  Each healthy subject will be imaged by the MIOCT system. There will be no surgery or intervention on these healthy volunteer subjects. We anticipate that a portion of the volunteer subjects would have repeat imaging (e.g. for reproducibility testing).
  Interventions: Device: Microscope integrated optical coherence tomography
- Surgeons as research subjects: Duke Eye Center surgical trainees (residents and fellows), attending surgeons, and surgeons from other medical institutions will be enrolled as subjects as we will test their performance with and without microscope integrated optical coherence tomography and with and without advances in 4D MIOCT in model surgeries in the research wet lab to better understand the utility of specific aspects and of this next generation MIOCT as a whole for specific anterior segment and retinal surgical tasks.
  Interventions: Device: Microscope integrated optical coherence tomography
- Surgical patients: Adult and minor (> 4 months of age) surgical patients will be enrolled to evaluate and obtain multiple images from the microscope integrated optical coherence tomography system during clinically indicated vitreoretinal and anterior segment surgical procedures.
  Interventions: Device: Microscope integrated optical coherence tomography

INTERVENTIONS:
Device: Microscope integrated optical coherence tomography — This is translational study in which subjects will either be imaged with a microscope integrated optical coherence tomography (MIOCT) system or they will use MIOCT during surgical procedures. OCT systems are optical imaging technology that allow non-contact imaging of the microanatomy of the retina, cornea, optic nerve head and retinal blood vessels. The MIOCT has been integrated into the surgical microscope used in retinal and anterior segment surgeries so it does not touch the eye. Unlike visible light from many examination devices, the infrared OCT beam is barely visible to the human eye as it sweeps across the retina. Thus the patient is not disturbed by the light.
  Other Names: MIOCT

SUMMARY:
The overall five-year goals of the project are to develop novel technology to provide actionable new information through provision of live volumetric imaging during surgery, improving surgical practice and outcomes. The investigators believe this technology will enable novel ophthalmic and other microsurgeries not possible due to current limitations in surgical visualization.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy controls: Healthy eyes without known disease: refractive error including myopia and non-significant cataract is allowed. For selected testing pseudophakia is allowed.
2. Surgeons as research subjects: Adult (≥18 years old)
3. Surgical patients (vitreoretinal surgery): Patients undergoing examination under anesthesia or surgery for vitreoretinal diseases
4. Surgical patients (anterior segment surgery-glaucoma, ocular surface or strabismus requiring extraocular muscle surgery): Include both adults and children. Patient undergoing primary, elective minimally invasive glaucoma surgery, ocular surface surgery, or strabismus surgery.

Exclusion Criteria:

1. Healthy controls: Any ocular disease that restricts the ability to perform OCT scanning. Conflict of interest with investigators/study personnel, e.g. a student in the lab of an investigator.
2. Surgeons as research subjects: no specific exclusion criteria.
3. Surgical patients (vitreoretinal surgery): Neonates (< 4 weeks of age) and patients with any ocular disease that restricts the ability to perform OCT scanning.
4. Surgical patients (anterior segment surgery-corneal and cataract diseases): Pediatric patients: The cornea and cataract surgery studies will be restricted to adults (≥ 18 years). Children do not have cataract surgery typically by residents and therefore would not fit our study design. Similarly pediatric corneal transplants are very rare.

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 262 subjects enrolled in 3 groups as follows:
  1. Healthy Controls: 50 subjects
  2. Surgeons as research subjects performing randomized testing in wet lab: 22 subjects
  3. Surgical patients as research subjects for application to ocular vitreoretinal and anterior segment surgery: 190 subjects
Sampling Method: Probability Sample
Enrollment: 262 (Estimated)
Dates: Start 2018-09-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Retinal and/or corneal microscope integrated optical coherence tomography image capture | Year 1
  Ability to capture images
Quality of retinal and/or corneal microscope integrated optical coherence tomography image capture | Year 1
  Quality of MIOCT images scored based on standard microanatomy and ability to detect presence or absence of ocular pathologies based on review by a masked grader.
Retinal vascular flow on optical coherence tomography angiography (OCTA) versus fluorescein angiography | Year 1
  Cross correlation of ability to capture vessels and vessel pathology between OCTA and fluorescein angiographic images.
Assessment of change in pattern of ocular vascular flow before and after standard clinical surgical steps. | Year 1
  Presence or absence of change in ocular morphology in pattern of vascular flow compared to prior to surgical steps
Assessment of change in ocular morphology before and after standard surgical steps | Year 1
  Presence or absence of change in ocular morphology before and after standard surgical steps
Estimate of subretinal fluid volume before and after surgery for retinal detachment based on surgical view versus based on OCT output | Year 1
  Volume estimates from surgeons analyzed relative to the postoperative calculated volume from the intraoperative MIOCT

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Toth, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No